CLINICAL TRIAL: NCT01855191
Title: Standardized Data Collection (SDC) for Lung Cancer Patients Treated With Curative Primary or Postoperative Radiotherapy or Chemoradiation (SDC Lung).
Brief Title: SDC for Lung Cancer Patients Treated With Curative Primary or Postoperative Radiotherapy or Chemoradiation
Acronym: SDC lung
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: SDC Lung
Record Dates: First submitted 2013-03-26; First posted 2013-05-16 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard
- Standard + saliva collection

SUMMARY:
Introducing standardized data collection (SDC) for lung cancer patients to improve the performance of the prediction models.

DETAILED DESCRIPTION:
All patients planned for curative primary or postoperative radiotherapy can be included. Patients will be treated according to the institutional protocol. It is optional to collect a saliva sample for genetic profiling.

Follow up at five time points:

* 2 weeks after RT
* 3 months after RT
* 6 months after RT
* 12 months after RT
* 24 months after RT

At these time points, toxicity will be assessed. In addition, patients will receive a short questionnaire by mail at eight time points.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for curatively intended radiotherapy or postoperative radiotherapy
* Recurrent disease

Exclusion Criteria:

* All patients planned for palliative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients planned for curatively intended radiotherapy or postoperative radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 864 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Two-year survival rate | 24 months after RT

SECONDARY OUTCOMES:
Change in dyspnea | during 24 months after RT
Change in cough | During 24 months after RT
Change in dysphagia | During 24 months after RT
Patient-rated generic quality of life | During 24 months after RT
  Measured by Euroqol questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD., PhD., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands